CLINICAL TRIAL: NCT02240394
Title: TCD Detection of Ophthalmic Artery Blood Flow Velocity Prediction Feasibility Study of Intracranial Pressure
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Xueming Wang, Chief Physician, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Other Study IDs: Shanghai6thPeoplesH
Record Dates: First submitted 2014-09-03; First posted 2014-09-15 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Traumatic Brain Injury; Cerebral Hemorrhage; Increased Intracranial Pressure
Keywords: TCD Traumatic brain injury increased intracranial pressure
MeSH Terms: conditions — Brain Injuries, Traumatic; Cerebral Hemorrhage; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Increased intracranial pressure is a cause of disease progression in patients with brain disease, a common cause of poor prognosis. Intracranial pressure monitoring is the observation of the disease, treatment, evaluation and important way to improve the prognosis. Non-invasive intracranial pressure monitoring can be used to stroke, intracranial hemorrhage, brain trauma, encephalitis and other patients. Ophthalmic artery originated from the internal carotid artery, the optic canal into the orbit, the entire process can be divided into intracranial optic tube segment and orbital segment. investigators' preliminary experiments show that when intracranial pressure, intracranial ophthalmic artery segment velocity increases with increasing velocity difference orbital segment. Accordingly, the investigators speculate, may be judged by the level of intracranial pressure intracranial and orbital velocity difference between the ophthalmic artery segment, and accordingly calculate the specific values of intracranial pressure. The investigators will collect brain trauma surgery, performed invasive intracranial pressure monitoring cases, the use of transcranial Doppler ultrasound velocity and different segments of the ophthalmic artery pulsatility index, the invasive intracranial pressure and comparing the measured values to calculate the the critical value of the ophthalmic artery segment intraorbital and intracranial velocity difference when intracranial pressure, thus fitting Based on projections of mathematical formulas intracranial pressure. This study will provide a non-invasive intracranial pressure monitor new approach.

DETAILED DESCRIPTION:
2014/08/28

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years of age (including 18 and 75 years), gender, ethnic limitation;
2. have been carried out invasive intracranial pressure monitoring;
3. the patient or his agent informed consent. -

Exclusion Criteria:

1. the patient does not fit, measured by TCD can not be completed;
2. TCD failed to detect the satisfaction of the ophthalmic artery flow signals were;
3. patients with ocular trauma or a history of intraocular pressure -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Traumatic brain injury patients has been in patients with invasive intracranial pressure monitoring
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Ophthalmic artery blood flow rate changes associated with intracranial pressure | "up to 6 months"

SECONDARY OUTCOMES:
the change of the Ophthalmic artery peak sistolic velocity associated with intracranial pressure | "up to 6 months"

OTHER OUTCOMES:
the change of the Ophthalmic artery end diastolic velocity associated with intracranial pressure | "up to 6 months"

CONTACTS AND LOCATIONS:
Overall Officials: Wang X Ming, Dr., Principal Investigator — World Health Organization
Locations (1):
- NCU, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Ragauskas A, Matijosaitis V, Zakelis R, Petrikonis K, Rastenyte D, Piper I, Daubaris G. Clinical assessment of noninvasive intracranial pressure absolute value measurement method. Neurology. 2012 May 22;78(21):1684-91. doi: 10.1212/WNL.0b013e3182574f50. Epub 2012 May 9. PMID 22573638